CLINICAL TRIAL: NCT01150760
Title: Comparison of Clinical Outcomes in Bowel Resection Patients Receiving Alvimopan vs. Patients Not Receiving Alvimopan in the Premier Perspective/Care Science Database
Brief Title: Clinical Outcomes After Bowel Resection in Patients Receiving Alvimopan Versus Patients Not Receiving Alvimopan in the Premier Perspective Database
Status: Completed | Type: Observational
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: Premier clinical outcomes
Record Dates: First submitted 2010-06-23; First posted 2010-06-25 (Estimated); Results first posted 2010-09-08 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2010-09

CONDITIONS: Ileus
Keywords: GI recovery after bowel resection; morbidity after bowel resection; mortality; readmission; length of stay
MeSH Terms: conditions — Ileus | interventions — alvimopan

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Alvimopan Users
  Interventions: Drug: Alvimopan
- Matched controls

INTERVENTIONS:
Drug: Alvimopan — At least 1 dose of alvimopan 12 mg during the hospitalization for bowel resection
  Other Names: Entereg
  Groups: Alvimopan Users

SUMMARY:
Alvimopan is the first and currently the only FDA-approved therapy for acceleration of the time to upper and lower gastrointestinal (GI) recovery following partial large or small bowel resection surgery with primary anastomosis.

The primary objective of this retrospective observational trial is to assess postoperative morbidity and mortality as reported during the index hospitalization for bowel resection and 15/30-day readmissions of alvimopan vs. non-alvimopan matched patients in the combined Premier/Care Science database(a large medical claims database).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years at discharge
* Medical claim with an ICD-9-CM procedure code for a primary procedure (identified at position 1 or 2 involving large or small segmental bowel resection with primary anastomosis
* Discharged within the study dates
* Surgery at a participating Premier/Care Sciences hospital

Exclusion Criteria:

* Had a diverting ostomy without a primary anastomosis during the index hospitalization
* Had a trauma diagnosis
* Had bowel resections performed on more than 1 day during index hospitalization (this includes cases where a bowel resection and intestinal anastomosis were performed on different days during the index hospitalization)
* Had an excluded non-bowel resection surgical code (i.e., code for a major non-BR surgical procedure [eg., nephroureterectomy, total joint replacement] in position 1 or 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective cohort study using the medical claims Premier/Care Science database. The study time frame was from January 1, 2009 through December 31, 2009.
Sampling Method: Probability Sample
Enrollment: 7050 (Actual)
Dates: Start 2010-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Techner, DPM, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (1):
- Premier database, Charlotte, North Carolina, United States

REFERENCES:
- [Derived] Delaney CP, Craver C, Gibbons MM, Rachfal AW, VandePol CJ, Cook SF, Poston SA, Calloway M, Techner L. Evaluation of clinical outcomes with alvimopan in clinical practice: a national matched-cohort study in patients undergoing bowel resection. Ann Surg. 2012 Apr;255(4):731-8. doi: 10.1097/SLA.0b013e31824a36cc. PMID 22388106

RESULTS

PARTICIPANT FLOW:
Groups:
- Alvimopan Users: Oral alvimopan 12 mg (dosing recommendation = once preoperatively then twice daily postoperatively for up to 15 in-hospital doses)
- Matched Controls: Each alvimopan patient was exact-matched (surgical procedure, surgeon specialty) and propensity score-matched (baseline characteristics) to a bowel resection patient who did not receive alvimopan
Period: Overall Study
Arm/Group | Alvimopan Users | Matched Controls
Started | 3525 | 3525
Completed | 3525 | 3525
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alvimopan Users | Matched Controls | Total
Number analyzed (Participants) | 3525 | 3525 | 7050
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (14.1) | 61.8 (14.7) | 61.9 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1847 | 1872 | 3719
  Male | 1678 | 1653 | 3331
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 331 | 368 | 699
  White | 2675 | 2543 | 5218
  Other | 519 | 614 | 1133
Procedure type [Number; unit: Participants] — Category of bowel resection that patients underwent during their hospitalization
  Participants
    Laparoscopic colon or rectal resection | 1427 | 1427 | 2854
    Open colon or rectal resection | 1171 | 1171 | 2342
    Laparoscopic or open colon or rectal resection | 424 | 424 | 848
    Laparoscopic or open small bowel resection | 181 | 181 | 362
    Laparoscopic or open ostomy takedown, bypass,other | 322 | 322 | 644
Surgeon type [Number; unit: Participants] — The type of surgeon that performed the patient's bowel resection during their hospitalization
  Participants
    General surgeon | 1809 | 1809 | 3618
    Colorectal surgeon | 1357 | 1357 | 2714
    Other | 359 | 359 | 718

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Died
Description: All-cause
Time Frame: Participants were followed up until their hospital discharge after bowel resection
Population: Intent-to-treat population (Included patients who meet all base population, inclusion and exclusion criteria, and had at least 1 administration of alvimopan [for the alvimopan cohort] during their hospitalization)
Measure: Number; unit: Percent of participants
Arm/Group | Alvimopan Users | Matched Controls
Number analyzed (Participants) | 3525 | 3525
Percent of participants | 0.4 | 1.0
Statistical Analysis 1: Comparison: Alvimopan Users vs Matched Controls; Test type: Superiority or Other; p = 0.0007, Chi-squared; Mean Difference (Net) = -0.6

2. Primary Outcome: Percentage of Patients With Reported In-hospital Postoperative Gastrointestinal (GI) Morbidity
Description: GI morbidity will be identified using International Classification of Disease 9th Edition Clinical Modification (ICD-9-CM) diagnosis and procedure codes for paralytic ileus, flatulence, eructation, gas pain, insertion of a nasogastric tube, total parenteral nutrition, peripheral parenteral nutrition, digestive symptom complications, diarrhea following GI surgery, intestinal obstruction, abdominal pain, peritoneal adhesions, unspecified protein-calorie malnutrition, parenteral infusion of concentrated nutritional substances, or enteral infusion of concentrated nutritional substances.
Time Frame: Participants were followed up until their hospital discharge after bowel resection
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | Alvimopan Users | Matched Controls
Number analyzed (Participants) | 3525 | 3525
Percent of participants | 29.8 | 35.7
Statistical Analysis 1: Comparison: Alvimopan Users vs Matched Controls; Test type: Superiority or Other; p < 0.0001, Chi-squared; Mean Difference (Net) = -5.9

3. Primary Outcome: Percentage of Patients With In-hospital Cardiovascular Morbidity
Description: Cardiovascular morbidity was identified using ICD-9-CM diagnosis and procedure codes for myocardial infarction; other ischemic events; congestive heart failure and shock; arrhythmias; or other cardiovascular events (cardiac complications, peripheral vascular complications).
Time Frame: Participants were followed up until their hospital discharge after bowel resection
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | Alvimopan Users | Matched Controls
Number analyzed (Participants) | 3525 | 3525
Percent of participants | 19.4 | 24.0
Statistical Analysis 1: Comparison: Alvimopan Users vs Matched Controls; Test type: Superiority or Other; p = 0.0001, Chi-squared; Mean Difference (Net) = -4.6

4. Primary Outcome: Percentage of Patients With In-hospital Cerebrovascular Morbidity
Description: Cerebrovascular morbidity was identified using ICD-9-CM diagnosis and procedure codes for ischemic, thrombotic, embolic or hemorrhagic cerebrovascular accidents; acute but ill-defined cerebrovascular disease; transient cerebral ischemia; syncope; or postoperative cerebrovascular accident.
Time Frame: Participants were followed up until their hospital discharge after bowel resection
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | Alvimopan Users | Matched Controls
Number analyzed (Participants) | 3525 | 3525
Percent of participants | 0.2 | 0.5
Statistical Analysis 1: Comparison: Alvimopan Users vs Matched Controls; Test type: Superiority or Other; p = 0.1022, Chi-squared; Mean Difference (Net) = -0.3

5. Primary Outcome: Percentage of Patients With In-hospital Pulmonary Morbidity
Description: Pulmonary morbidity was identified using ICD-9-CM diagnosis and procedure codes for pneumonia; infectious pneumonia; respiratory complications, pulmonary collapse; acute respiratory failure or edema; pulmonary congestion and hypostasis; pulmonary/respiratory insufficiency after trauma and/or surgery; dyspnea; or respiratory arrest; transfusion related acute lung injury.
Time Frame: Participants were followed up until their hospital discharge after bowel resection
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | Alvimopan Users | Matched Controls
Number analyzed (Participants) | 3525 | 3525
Percent of participants | 7.3 | 10.5
Statistical Analysis 1: Comparison: Alvimopan Users vs Matched Controls; Test type: Superiority or Other; p < 0.0001, Chi-squared; Mean Difference (Net) = -3.2

6. Secondary Outcome: Postoperative Length of Hospital Stay
Description: Calendar day of discharge - calendar day of surgery = postoperative length of stay
Time Frame: Measured from the day after bowel resection to the day of hospital discharge
Population: Modified intent-to-treat (included patients who met all base population, inclusion and exclusion criteria, received ≥ 3 and ≤ 15 doses of alvimopan [for alvimopan cohort] during the patient's hospitalization, and received parenteral opioid on ≥ 1 postoperative day)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Alvimopan Users | Matched Controls
Number analyzed (Participants) | 2323 | 2323
Days | 5.3 (3.1) | 6.4 (4.8)
Statistical Analysis 1: Comparison: Alvimopan Users vs Matched Controls; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -1.1

7. Primary Outcome: Percentage of Patients With In-hospital Infection Morbidity
Description: Infection morbidity was identified using ICD-9-CM diagnosis and procedure codes for infection due to central venous catheter; abscess of intestine; peritoneal abscess; sepsis or severe sepsis; infection due to vascular device, implant and graft; urinary tract infection; disruption of internal or external surgical wound; persistent postoperative fistula; or postoperative infection.
Time Frame: Participants were followed up until their hospital discharge after bowel resection
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | Alvimopan Users | Matched Controls
Number analyzed (Participants) | 3525 | 3525
Percent of participants | 9.2 | 11.5
Statistical Analysis 1: Comparison: Alvimopan Users vs Matched Controls; Test type: Superiority or Other; p = 0.0012, Chi-squared; Mean Difference (Net) = -2.3

8. Primary Outcome: Percentage of Patients With In-hospital Thromboembolic Morbidity
Description: Thromboembolic morbidity was identified using ICD-9-CM diagnosis and procedure codes for pulmonary embolism and infarction; arterial embolism and thrombosis or thrombosis of the lower extremities; vascular disorders of the kidney; acute vascular insufficiency of the intestine; or venous thromboembolism.
Time Frame: Participants were followed up until their hospital discharge after bowel resection
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | Alvimopan Users | Matched Controls
Number analyzed (Participants) | 3525 | 3525
Percent of participants | 1.2 | 2.1
Statistical Analysis 1: Comparison: Alvimopan Users vs Matched Controls; Test type: Superiority or Other; p = 0.0030, Chi-squared; Mean Difference (Net) = -0.9

9. Primary Outcome: Percentage of Patients With In-hospital Other Morbidity
Description: Other morbidity was identified using ICD-9-CM diagnosis and procedure codes for disruption of wound, decubitus ulcer, or postoperative complications not elsewhere classified.
Time Frame: Participants were followed up until their hospital discharge after bowel resection
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | Alvimopan Users | Matched Controls
Number analyzed (Participants) | 3525 | 3525
Percent of participants | 0.6 | 0.7
Statistical Analysis 1: Comparison: Alvimopan Users vs Matched Controls; Test type: Superiority or Other; p = 0.7637, Chi-squared; Mean Difference (Net) = -0.1

10. Primary Outcome: Percentage of Patients Who Were Readmitted Within 15 Days of Discharge
Time Frame: Within 15 days of discharge from hospitalization for bowel resection
Population: Intent-to-treat population (included patients who met all base population, inclusion and exclusion criteria, and had at least 1 administration of alvimopan [for the alvimopan cohort] during the patient's hospitalization)
Measure: Number; unit: Percent of partcipants
Arm/Group | Alvimopan Users | Matched Controls
Number analyzed (Participants) | 3525 | 3525
Percent of partcipants | 7.4 | 8.7
Statistical Analysis 1: Comparison: Alvimopan Users vs Matched Controls; Test type: Superiority or Other; p = 0.0402, Chi-squared; Mean Difference (Net) = -1.3

11. Primary Outcome: Percentage of Patients Who Were Readmitted Between 16 and 30 Days After Discharge
Time Frame: Between 16-30 days after hospital discharge after bowel resection
Population: as for outcome 10
Measure: Number; unit: Percent of participants
Arm/Group | Alvimopan Users | Matched Controls
Number analyzed (Participants) | 3525 | 3525
Percent of participants | 1.9 | 2.5
Statistical Analysis 1: Comparison: Alvimopan Users vs Matched Controls; Test type: Superiority or Other; p = 0.0755, Chi-squared; Mean Difference (Net) = -0.6

12. Primary Outcome: Percentage of Patients Who Were Readmitted Within 30 Days of Discharge
Time Frame: Between 0-30 days after hospital discharge after bowel resection
Population: as for outcome 10
Measure: Number; unit: Percent of participants
Arm/Group | Alvimopan Users | Matched Controls
Number analyzed (Participants) | 3525 | 3525
Percent of participants | 9.3 | 11.2
Statistical Analysis 1: Comparison: Alvimopan Users vs Matched Controls; Test type: Superiority or Other; p = 0.0532, Chi-squared; Mean Difference (Net) = -1.9

13. Primary Outcome: Percentage of Patients Discharged to Various Locations
Description: Location of discharge for patients who were admitted to the hospital for their bowel resection from home
Time Frame: Hospital discharge after bowel resection
Population: as for outcome 10
Measure: Number; unit: Percent of participants
Arm/Group | Alvimopan Users | Matched Controls
Number analyzed (Participants) | 3525 | 3525
Percent of participants
  Health care facility | 7.9 | 13.8
  Home | 87.5 | 80.7
Statistical Analysis 1: Comparison: Alvimopan Users vs Matched Controls; Test type: Superiority or Other; p < 0.0001, Chi-squared

14. Primary Outcome: Intensive Care Unit Length of Stay
Time Frame: Participants were followed up until their hospital discharge after bowel resection
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Alvimopan Users | Matched Controls
Number analyzed (Participants) | 3525 | 3525
Days | 0.3 (1.4) | 0.6 (2.4)
Statistical Analysis 1: Comparison: Alvimopan Users vs Matched Controls; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -0.3

ADVERSE EVENTS:
Description: Adverse events were not collected in this retrospective observational study.
Arm/Group | Alvimopan Users | Matched Controls
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No